CLINICAL TRIAL: NCT05731882
Title: First in Man Study to Evaluate Safety and Efficacy of Left Atrial Appendage Pulsed Field Ablation Occluder for Simultaneous Pulsed Field Ablation and Mechanical Closure of the Left Atrial Appendage in Patients With Nonvalvular Atrial Fibrillation
Brief Title: First in Man Study of Left Atrial Appendage Pulsed Field Ablation Occluder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Dinova EP Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-SeaLA FIM 01
Record Dates: First submitted 2023-01-30; First posted 2023-02-16 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Nonvalvular Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Catheter ablation+E-SeaLATM (Experimental)
  Interventions: Device: E-SeaLA, CardioPulse PFA system

INTERVENTIONS:
Device: E-SeaLA, CardioPulse PFA system — First, pulmonary vein isolation(PVI) was performed with the novel hex spline PFA ablation catheter( CardioPulseTM PFA system, Hangzhou Dinova EP Technology Co., Ltd), then, pulsed field ablation and mechanical closure of the left atrial appendage were achieved by E-SeaLATM(Hangzhou Dinova EP Technology Co., Ltd) implantation.

SUMMARY:
This is the first in man study of E-SeaLATM developed and manufactured by Hangzhou Dinova EP Technology Co., Ltd, which can achieve pulsed field ablation and mechanical closure of the Left Atrial Appendage simultaneously, this study aims to initially verify the safety and efficacy of the device.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the patient is 18~80 years old;
2. patients diagnosed with non-valvular atrial fibrillation (at least 1 episode of atrial fibrillation recorded on ECG or Holter in the 12 months prior to enrollment);
3. CHA2DS2-VASC score: male≥ 2, female≥ 3;
4. patients are not suitable for long-term oral anticoagulant therapy (any of the following): (1) not suitable for long-term standardized anticoagulation therapy; (2) stroke or embolism still occurs on the basis of long-term standardized anticoagulation therapy; (3) HAS-BLED score≥ 3 points; (4) need to be treated with antiplatelet drugs; (5) unwillingness to undergo long-term anticoagulant therapy;
5. Be able to understand the purpose of the study, voluntarily participate in the study, sign the informed consent form by the subject himself or her legal representative, and be willing to complete the follow-up in accordance with the requirements of the program.

Exclusion Criteria:

1. Atrial fibrillation secondary to electrolyte imbalances, thyroid disease or other reversible factors;
2. Left atrial appendage depth < 15mm, left atrial appendage anchor area < 10mm or >33mm;
3. Left atrial diameter≥ 65mm;
4. Imaging examination shows left atrium or left atrial appendage thrombosis;
5. Severe structural heart disease (such as moderate to severe aortic valve, mitral stenosis or regurgitation);
6. Left ventricular ejection fraction <35%, or New York College of Cardiology class III or IV;
7. Refractory hypertension (blood pressure persists > 180/110mmHg after treatment);
8. Patients with previous patent foramen ovale closure, atrial septal defect closure or repair;
9. Patients with previous left atrial appendage occlusion or left atrial appendage closure;
10. Patients with previous valve repair, prosthetic valve implantation or replacement;
11. Patients who have implanted devices such as implantable cardioverter defibrillator(ICD), cardiac resynchronization therapy(CRT) or pacemaker or have an implantation plan within 12 months after procedure;
12. Patients with clinically symptomatic carotid artery stenosis, or patients who have undergone carotid stenting or carotid endarterectomy in the past 6 months;
13. Patients with a history of myocardial infarction in the past 6 months, or who have undergone coronary artery bypass grafting or percutaneous coronary intervention;
14. Recorded thromboembolic events (including transient ischemic attack) in the past 30 days;
15. Serum creatinine greater than 2 times the upper limit of normal, or history of renal dialysis;
16. Acute systemic infection;
17. Severe lung disease, pulmonary hypertension or any lung disease involving abnormal blood gases or severe breathing difficulties;
18. Presence of wall thrombosis, tumors or other abnormalities that interfere with vascular puncture or catheter operation;
19. Female patients who are pregnant, lactating, or unable to use contraception during the study;
20. patients have participated in clinical trials of other drugs or devices during the same period;
21. patient's life expectancy is less than 12 months;
22. Abnormalities or diseases that the investigator believes should be excluded from the scope of enrollment in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-07-17 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | immediately after the procedure
  Technical success means that the pulmonary vein and left atrial appendage(LAA) remain electrical isolation 20 minutes after ablation, and the per-device leaks≤ 3 mm after E-SeaLA LAA pulsed field ablation(PFA) occluder implantation.
The incidence of major adverse events (MAEs) related to devices or procedures 3 months after procedure | within 3 months after procedure
  MAE includes death, myocardial infarction, stroke or transient ischemic attack (TIA), pulmonary vein stenosis, phrenic nerve palsy, systemic embolism, pericarditis, pericardial effusion/cardiac tamponade, atrial esophageal fistula, severe vascular access complications, device migration, and device embolization.

SECONDARY OUTCOMES:
Ablation efficiency including total procedure time, catheter dwell time, total ablation time and total X-ray exposure time | immediately after the procedure
  Total procedure time (defined as the total time from initial femoral venipuncture to final catheter removal), catheter dwell time (time between the pulsed field ablation catheter entering the left atrium and its withdrawal from the left atrium), total ablation time (including total PVI ablation time, total LAA ablation time), total X-ray exposure time (the total time of X-ray imaging of the catheter).
Left atrial appendage closure rate 12 months after procedure | within 12 months after procedure
  after occlusion device implantation, no forward or reverse blood flow through the occluder confirmed by ultrasound, residual forward or reverse blood flow at the edge of the occluder ≤3mm, peri-device leaks ≥grade 3)
Incidence of ischemic stroke within 12 months after procedure (event/patient-year). | within 12 months after procedure
  Ischemic stroke refers to the loss of neurological function caused by transient ischemic attack, cerebral thrombosis or cerebral embolism caused by the lesions of the brain itself and/or systemic blood circulation disorders leading to cerebral blood supply disorders. Ischemic stroke is defined as a modified Rankin score (mRS) ≥2 90 days after stroke onset.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - General Hospital of Northern Theater Command, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: Undecided